CLINICAL TRIAL: NCT03566667
Title: Beta-blockeRs tO patieNts With CHronIc Obstructive puLmonary diseasE
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Ole Frobert, MD, PhD (Other)
Responsible Party: Sponsor-Investigator, Ole Frobert, MD, PhD, Professor, Region Örebro County
Organization: Region Örebro County (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BRONCHIOLE-2017
Record Dates: First submitted 2018-06-12; First posted 2018-06-25 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-04

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Beta-blockers
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Metoprolol; Standard of Care

STUDY DESIGN:
Intervention Model Description: Pragmatic randomized controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Metoprolol (Active Comparator): Metoprolol at an aimed dose of 100 mg in addition to usual standard care
  Interventions: Drug: Metoprolol
- Standard care (Other): Usual standard care
  Interventions: Drug: Standard care

INTERVENTIONS:
Drug: Metoprolol — Betablocker
  Arms: Metoprolol
Drug: Standard care — Standard care
  Other Names: Usual standard care
  Arms: Standard care

SUMMARY:
Background: In patients with chronic obstructive pulmonary disease (COPD) and concomitant cardiovascular conditions cardio-selective beta-blockers reduce mortality and can be used without significant negative effects on lung function or respiratory symptoms. Observational studies indicate that beta-blocker therapy in COPD even without overt cardiovascular disease, is associated with reduced risk for mortality and COPD exacerbations.

Aim: The overall purpose of our study is to examine the benefit of general beta-blocker therapy on important patient-oriented measures in chronic obstructive pulmonary disease (COPD). Our primary hypothesis that treatment with beta-blockers in patients with COPD and no comorbid heart disease at baseline can prevent a Composite measure of hospitalizations due to cardiovascular diseases, COPD exacerbations and death.

Population: 1700 patients with C OPD. Inclusion criteria are FEV1/FVC < 70, age >40 years and sinus rhythm 50-120/min. Exclusion criteria include hypersensitivity against metoprolol, atrioventricular (AV) block II or II or sick sinus syndrome without pacemaker, atrial fibrillation or flutter, clinical signs of or previously known cardiovascular disease, systolic blood pressure < 90, severe asthma, present beta-blocker therapy or ongoing COPD exacerbation.

Intervention: Metoprolol at a target dose of 100 mg in addition to standard COPD care.

Control: No placebo control. Randomized, pragmatic un-blinded controlled study where the control Group receives standard COPD care.

Outcome: The primary outcome is a composite measure of all-cause mortality, C OPD exacerbations, and cardiovascular events after one year. Endpoint data from Swedish national registries and clinical follow-up.

Importance: Beta-blocker treatment to attenuate morbidity in patients with COPD could have great clinical and social importance at a low cost.

DETAILED DESCRIPTION:
Purpose and aims

The overall purpose of our study is to examine the benefit of general beta-blocker therapy on important patient-oriented measures in chronic obstructive pulmonary disease (COPD). Our primary aim is to examine if treatment with beta-blockers in patients with COPD and no comorbid heart disease at baseline can prevent hospitalizations due to cardiovascular diseases, COPD exacerbations and death.

Background

In patients with chronic obstructive pulmonary disease (COPD) and concomitant cardiovascular conditions cardio-selective beta-blockers reduce mortality and can be used without significant negative effects on lung function or respiratory symptoms. Observational studies indicate that beta-blocker therapy in COPD even without overt cardiovascular disease, is associated with reduced risk for mortality and COPD exacerbations.

Research questions

Primary: Does treatment with metoprolol at an aimed dose of 100 mg in addition to standard care statistically significantly decrease the one year rate of a composite measure of death, COPD exacerbations or hospitalization due to a cardiovascular event, in patients with COPD and no cardiovascular disease at baseline? Secondary: Does treatment with metoprolol at an aimed dose of 100 mg in addition to standard care: -decrease the one year rate of a death (all-cause and cause-specific), in patients with COPD and no cardiovascular disease at baseline? -decrease the one year rate of exacerbations, in patients with COPD and no cardiovascular disease at baseline? -decrease the one year rate of hospitalization for myocardial infarction, angina pectoris, heart failure, atrial fibrillation or other forms of arrhythmia, stroke, transient ischemic attack (TIA) or cerebral hemorrhage in patients with COPD and no cardiovascular disease at baseline?

Study design

This is a randomized controlled clinical trial (RCCT) with a pragmatic approach, i.e. a study characterized by a minimized number of inclusion and exclusion criteria, a reduced number of follow-up visits, a reduced complexity at the visits, and an intervention that is additional to standard care but with no placebo control (Figure 1). Invitation letters are sent to all patients, managed at the Department of Respiratory Medicine at Orebro University Hospital or primary health care centers in Region Orebro County, with a doctor´s diagnosis of COPD, no International Classification of Diseases (ICD) codes for cardiovascular diseases and no present beta-blocker therapy.

Inclusion and follow-up will take place at the Clinical Research Support Center in Orebro. In addition, several other Swedish centers for clinical trials have accepted to take part in the study.

The intervention with metoprolol at an aimed dose of 100 mg is prescribed electronically through the ordinary record system, and with financial burdening of the project unless the patient is already part of the high-cost protection for medication. A total of 1700 patients will be randomized to standard care or intervention.

Estimated sample size and statistical power

Sample size is calculated on the basis of: 1) an estimated overall 1-year risk of death of 1% in this mixed cohort of patients with various stages of COPD, 2) a 1-year risk for COPD exacerbations of 20% and 3) a 1-year risk of myocardial infarction, atrial fibrillation, other arrhythmias, heart failure, stroke, TIA or cerebral hemorrhage leading to hospitalization of 2%. The combined 1-year primary endpoint is estimated at 23% (expected survival probability of 0.77) for individuals randomized to usual standard care. With a 5% two-sided alpha level and statistical power set to 80%, 763 patients in each group (total n=1526) is needed to detect a 25% reduction of the primary endpoint in the beta blocker group, corresponding to a hazard ratio of 0.75. In order to control for dropouts and crossing from one group to the other 1700 patients will be included.

Statistical analysis plan

Analysis according to the intention-to-treat principle. Differences between groups in the time-to-event-end points will be assessed using the log-rank test, Kaplan-Meier methodology and Cox proportional hazard model. Differences between study groups will be assessed with unpaired t-tests on original scale or log scale as appropriate. Ordinal variables will be assessed with chi-2 test for trend or Mann-Whitney U test, and Pearson's chi-square test or Fisher's exact test will be used to test differences between proportions. Subgroup analyses will be carried out for patients with a resting heart rate of <80 vs. ≥80 beats per minute.

Randomization procedure and and study data base

Following written informed consent randomization is performed with a 1:1 allocation using the Smart Trial system web page. A study data base with all patients included in the study will be generated within the Smart-Trial system. The patients' identity will always be confidential.

Monitoring

In accordance with the principles of International Council for Harmonisation of Technical Requirements for Pharmaceuticals for Human Use - Good Clinical Practice (ICH-GCP), monitoring of the study will be arranged by the Sponsor and occur on site before, during and after the trail. During the study, monitors will have regular contacts with the study site to ensure that the study is conducted and documented properly in compliance with the protocol, Standard Operating Procedures (SOPs), ICH-GCP and applicable regulatory requirements.

The number of monitoring visits will occur throughout the trial. The main part of the monitoring will be centralized by regular checks of the data quality in the database. The monitors will review source documents for verification of consistency with the study data recorded in an electronic case report form (eCRF) according to risk based monitoring. Investigators and other responsible personnel must be available during the monitoring visits, possible audits and inspections and should devote sufficient time to these processes.

Ethical considerations

The study will be conducted in accordance with the protocol, applicable regulatory requirements such as and the ethical principles of the Declaration of Helsinki as adopted by the 18th World Medical Assembly in Helsinki, Finland, in 1964 and subsequent versions. The study is approved by the Regional Ethical Review Board of Uppsala, Sweden (DNr 2017-210B) and the Swedish Medical Products Agency (EudraCT no: 2017-001507-76).

Reporting procedures for Adverse Events (AE) and Serious Adverse Events (SAE)

Only AE and SAE that are not considered as signs and symptoms expected and related to the endpoints or known side effects from the study drug will be reported in this study. Events defined as endpoints in the study (e.g. all-cause death, (cardiovascular events requiring hospitalization or COPD exacerbations) will not be reported as AE. This means that other clinical signs and symptoms, which are reported by the patient and observed by the investigator, and in the opinion of the investigator are unexpected in relation to actual diagnosis, will be reported.

Suspected Unexpected Serious Adverse Event (SUSAR) reporting procedure

If the responsible investigator judges the SAE as being drug-related and unexpected (SUSAR) the event must be reported to the sponsor within one working day. SUSARs will be reported using the Council for International Organizations of Medical Sciences (CIOMS) form (http://www.cioms.ch/index.php/cioms-form-i) which will be sent to the Medical Products Agency, since sponsor is not able to report electronically to the EudraVigilance database. The sponsor is responsible for information to all involved investigators in the study.

Annual report

A safety report, including assessment of overall safety and all reported SUSARs will be submitted yearly to the Regulatory Authorities and if requested to the Ethics Committee.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of COPD confirmed by spirometry showing post bronchodilator value of Forced Expiratory Volume in one second (FEV1)//Forced Vital Capacity (FVC) < 70 according to the Global Initiative on Obstructive Pulmonary Disease (GOLD)
* ≥40 years of age
* Sinus rhythm ≥50/min and <120 at inclusion

Exclusion Criteria:

* Known hypersensitivity to metoprolol or related derivatives
* AV block II or III unless treated with a pacemaker
* Sinus bradycardia (resting heart rate <50/min)
* Sick sinus syndrome unless treated with a pacemaker
* Atrial fibrillation/flutter
* Clinical signs of or a previous diagnosis of heart failure, angina pectoris, myocardial infarction, cerebrovascular disease or critical peripheral ischemia
* Systolic blood pressure <90 mmHg
* Any tachy-arrythmias other than sinus rhythm
* Sinus tachycardia >120 / min
* Systolic blood pressure <90 mmHg
* Severe bronchial asthma
* Current beta-blocker treatment
* Inability to provide informed consent
* Age below 40 years
* Acute on-going exacerbation of COPD
* Previous randomization in the BRONCHIOLE trial
* Ongoing pregnancy (excluded by pregnancy test in fertile women)

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1713 (Actual)
Dates: Start 2018-06-12 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Mortality, exacerbations and cardiovascular events | One year
  A composite measure of all-cause mortality, COPD exacerbations and cardiovascular events after one year

SECONDARY OUTCOMES:
Mortality | One year
  All-cause mortality after one year
Exacerbations | One year
  Number of COPD exacerbations after one year
Cardiovascular events | One year
  Number of cardiovascular events after one year

CONTACTS AND LOCATIONS:
Overall Officials: Ole Fröbert, MD, PhD, Study Chair — Region Örebro County
Locations (1):
- University Hospital of Örebro, Örebro, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Short PM, Lipworth SI, Elder DH, Schembri S, Lipworth BJ. Effect of beta blockers in treatment of chronic obstructive pulmonary disease: a retrospective cohort study. BMJ. 2011 May 10;342:d2549. doi: 10.1136/bmj.d2549. PMID 21558357
- [Result] Salpeter S, Ormiston T, Salpeter E. Cardioselective beta-blockers for chronic obstructive pulmonary disease. Cochrane Database Syst Rev. 2005 Oct 19;2005(4):CD003566. doi: 10.1002/14651858.CD003566.pub2. PMID 16235327
- [Result] Dransfield MT, Rowe SM, Johnson JE, Bailey WC, Gerald LB. Use of beta blockers and the risk of death in hospitalised patients with acute exacerbations of COPD. Thorax. 2008 Apr;63(4):301-5. doi: 10.1136/thx.2007.081893. Epub 2007 Oct 19. PMID 17951276
- [Result] Rutten FH, Zuithoff NP, Hak E, Grobbee DE, Hoes AW. Beta-blockers may reduce mortality and risk of exacerbations in patients with chronic obstructive pulmonary disease. Arch Intern Med. 2010 May 24;170(10):880-7. doi: 10.1001/archinternmed.2010.112. PMID 20498416
- [Derived] Sundh J, Magnuson A, Montgomery S, Andell P, Rindler G, Frobert O; BRONCHIOLE investigators. Beta-blockeRs tO patieNts with CHronIc Obstructive puLmonary diseasE (BRONCHIOLE) - Study protocol from a randomized controlled trial. Trials. 2020 Jan 30;21(1):123. doi: 10.1186/s13063-019-3907-1. PMID 32000825